CLINICAL TRIAL: NCT06137014
Title: Reduction of Severity and Duration of Pediatric Gastroenteritis Through Amino Acid Fortified Oral Rehydration Therapy
Brief Title: Fortified Oral Rehydration Therapy for Pediatric Diarrhea
Acronym: fORT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Paul A Breslin (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor-Investigator, Paul A Breslin, Professor of Nutritional Sciences, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro2021002499
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Gastroenteritis
Keywords: Gastroenteritis; Intestinal Diseases; Pediatric Diseases; Diarrhea, Infantile
MeSH Terms: conditions — Gastroenteritis; Intestinal Diseases; Diarrhea, Infantile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amino acid-fortified oral rehydration therapy (Experimental): Participants will consume the amino acid-fortified oral rehydration therapy (fORT) according to the World Health Organization (WHO) Treatment Plan A for ORT administration:
  * Child under 24 months: 50 to 100 ml ORT after each loose stool (approximately 500 ml daily)
  * Child from 2 to 10 years: 100 to 200 ml ORT after each loose stool (approximately 1000 ml daily)
  Interventions: Drug: Fortified Oral Rehydration Therapy
- Standard of care oral rehydration therapy (Placebo Comparator): Participants will consume the standard of care oral rehydration therapy according to the WHO Treatment Plan A for ORT administration:
  * Child under 24 months: 50 to 100 ml after each loose stool (approximately 500 ml daily)
  * Child from 2 to 10 years: 100 to 200 ml after each loose stool (approximately 1000 ml daily)
  Interventions: Dietary Supplement: Standard of Care Oral Rehydration Therapy

INTERVENTIONS:
Drug: Fortified Oral Rehydration Therapy — Oral rehydration solution with reduced glucose and added amino acids.
  Other Names: FORT
  Arms: Amino acid-fortified oral rehydration therapy
Dietary Supplement: Standard of Care Oral Rehydration Therapy — Glucose-based oral rehydration therapy according to World Health Organization guidelines.
  Arms: Standard of care oral rehydration therapy

SUMMARY:
The goal of this clinical trial is to compare amino acid-fortified oral rehydration therapy (ORT) to the standard of care ORT in pediatric patients with acute gastroenteritis (AGE). The main questions it aims to answer are:

* can amino acid-fortified ORT reduce the duration and severity of AGE compared to standard of care ORT?
* can amino acid-fortified ORT increase the secretion of antimicrobial peptides in the gastrointestinal tract compared to standard of care ORT?

Participants will be assigned to the experimental treatment (amino acid-fortified ORT) or the standard of care ORT and their disease severity, duration, and stool antimicrobial peptide content.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 6 months and 5 years.
* Experiencing mild to moderate acute gastroenteritis for less than two (2) days before admission to Pediatric Emergency Department.
* Diarrhea presumed infectious

Exclusion Criteria:

* Severe gastroenteritis with moderate to severe dehydration
* Requiring inpatient care
* Requiring antibiotics
* Requiring IV rehydration
* History of chronic diarrhea
* Presenting with diarrhea for greater than 2 days prior to admission
* Allergy to any of the ingredients in the study products
* Inborn metabolic disorder of amino acids
* Receives post-pyloric feedings

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Daily Stool Frequency | Up to 14 days
  Number of bowel movements (BMs) per day (count)
Daily Stool Mass | Up to 14 days
  Total mass of stool per day from measured BMs in grams
Duration of Diarrhea | Up to 14 days
  Duration of diarrhea in hours from onset until 3 formed stools in a row

SECONDARY OUTCOMES:
Consumption of Study Intervention | Up to 14 days
  Mls of ORT or FORT consumed per day
Stool Consistency | Up to 14 days
  Stool consistency rated on the Bristol Stool Scale
Body Weight | Up to 14 days
  Weight of child each day of study in kg
Stool Human Beta-Defensin-2 Content | Up to 14 days
  Beta-defensin-2 measured from stool sample in ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Paul Breslin, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share all de-identified data upon request by other researchers upon submission of manuscripts to journals.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: These will be made available to researchers and editors upon submission of manuscripts to journals for a period of up to 7 years post publication.
Access Criteria: Qualified independent researchers with an academic interest in pediatric GI disease. These data will be provided following review and approval of a research proposal, statistical analysis plan, and execution of a data sharing plan.